CLINICAL TRIAL: NCT04997096
Title: Exercise as a Preventive Agent to Combat Immobility in Patients With Ovarian or Endometrial Cancers Receiving Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Christina Dieli-Conwright, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-299
Record Dates: First submitted 2021-08-04; First posted 2021-08-09 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Ovarian Cancer; Ovarian Carcinoma; Ovarian Cancer Stage IV; Ovarian Cancer Stage III; Ovarian Cancer Stage 3; Endometrial Cancer; Endometrial Cancer Stage
Keywords: Ovarian Cancer; Ovarian Carcinoma; Ovarian Cancer Stage IV; Ovarian Cancer Stage III; Ovarian Cancer Stage 3; Endometrial Cancer; Aerobic Exercise; Strength Training; Cardiovascular training
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Participants randomized to one of two groups with 2:1 ratio: exercise (n=20)
  - Aerobic and Resistance Exercise for 16 weeks
  Interventions: Other: Exercise
- Attention Control (Active Comparator): Participants randomized to one of two groups with attention control (n=10).
  -Attention Control for 16 weeks home-based stretching
  Interventions: Other: Attention Control

INTERVENTIONS:
Other: Exercise — 16-week, virtually supervised, technology-based, aerobic and resistance exercise program performed 3 days per week which starts at least 4 weeks after surgery
  Arms: Exercise
Other: Attention Control — Home-based stretching program consisting of one set of 4 static stretching exercises held for 30 seconds and performed 3 days/week. Participants will be shown how to use the booklet and instructed on how to complete the stretching exercises by an exercise trainer.
  Arms: Attention Control

SUMMARY:
The purpose of this research is to determine whether a 16-week virtually supervised aerobic and resistance exercise program is feasible in patients receiving first-line chemotherapy after surgery for ovarian or endometrial cancer and if it will improve lower extremity function (function of the legs), lessen chemotherapy-induced peripheral neuropathy (CIPN; numbness or tingling in the hands or feet), and if there is any effect on inflammatory blood markers (the level of a certain marker in the blood that is associated with inflammation; redness and swelling).

DETAILED DESCRIPTION:
This research study is a randomized controlled trial that will compare an exercise group to a control group on lower extremity function, CIPN, and inflammatory markers in ovarian or endometrial cancer patients undergoing first-line chemotherapy after surgery.

The names of the study interventions involved in this study are/is:

* Aerobic and resistance exercise; virtually supervised 16-week aerobic and resistance exercise performed at home via Zoom
* Attention control for 16 weeks, home-based stretching

The research study procedures include: screening for eligibility and study interventions including evaluations and follow up visits.

It is expected that about 30 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with stages III-IV ovarian or endometrial cancer
* Receiving first-line carboplatin and paclitaxel chemotherapy after surgery
* ≥18 years, children under the age of 18 will be excluded due to rarity of disease
* Physician's clearance to participate in moderate-vigorous intensity exercise
* Able to read, write, and understand English
* Ability to understand and the willingness to sign an informed consent document
* Willing to undergo two venous blood draws for the study

Exclusion Criteria:

* Pre-existing musculoskeletal, neurological, or cardiorespiratory conditions, as determined by the treating oncologist
* Participants with uncontrolled intercurrent illness, as determined by the treating oncologist
* Participants with psychiatric illness/social situations that would limit compliance with study requirements, as determined by the treating oncologist
* Participants who have received prior chemotherapy for cancer treatment (e.g. taxanes for breast cancer)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-02 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients completing the exercise intervention sessions. | 16 Weeks
  The feasibility of the 16-week exercise intervention is defined as the proportion of patients completing the exercise intervention sessions. The analysis population will be the eligible patients who are assigned to the intervention group (N=20). The investigators will estimate the proportion and corresponding 95% exact confidence interval (CI).99 The Investigators expect that the proportion is 70% or higher
Enrollment Rate | 16 Weeks
  The enrollment rate is defined as the proportion of patients who participate in the study among those patients who are approached for the enrollment.

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPPB)-Lower Extremity Function | 16 Weeks
  Short Physical Performance Battery (SPPB), an objective measure of lower-extremity function based on three timed tests of standing balance, walking speed, and chair stand tests, which in older adults is predictive of disability, nursing home admission, and all-cause mortality
Change in 6-minute walk distance | 16 weeks
  Aerobic fitness will be assessed by the 6-minute walk test (6MWT). The 6MWT has been administered in cancer survivors and has a reliability coefficient of 0.93 when tested in cancer survivors. Participants will be instructed to walk as quickly as possible without running on an indoor pre-measured walkway for 6 minutes
PROMIS- Physical function | 16 Weeks
  Physical function will be assessed using the Patient Reported Outcome Measure Information System (PROMIS) Physical Function-10 scale.
Number of Participants with Treatment Related Adverse Events | 16 Weeks
  NCI Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Dieli-Conwright, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu